CLINICAL TRIAL: NCT03578653
Title: Merging Yoga and Occupational Therapy for Parkinson Disease: Phase 2
Acronym: MY-OT for PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17-7398H
Record Dates: First submitted 2018-06-13; First posted 2018-07-06 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Merging Yoga and Occupational Therapy for Parkinson disease (Experimental): The group participates in three assessment periods: August, October, and December. Then in October-December the group will receive group occupational therapy and recommended community adaptive yoga programming 2x/week for 8 weeks.
  Interventions: Behavioral: Merging Yoga and Occupational Therapy for Parkinson disease

INTERVENTIONS:
Behavioral: Merging Yoga and Occupational Therapy for Parkinson disease — The group occupational therapy portion focuses on lecture, group discussion, and activities to reduce fall risk. The yoga program is part of an ongoing community yoga program specifically designed for people with Parkinson disease.

SUMMARY:
The full program is focused on identifying and reducing risk factors surrounding falls. Based on previous research, we believe that occupational therapy group classes and adaptive yoga are an ideal pairing to reduce fall risk. The occupational therapy sessions will consist of lecture, group discussion, and activities designed to target biological, behavioral, environmental, and socioeconomic factors that contribute to fall risk specifically for people with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a diagnosis of Parkinson's disease OR their care partners
* Individuals who read and understand English
* Individuals who can stand with or without an assistive device
* People who are willing to commit to yoga practice 2x/week for 8 weeks and pay $5/class through Raintree Athletic Club (Scholarships are available if needed!)
* People who are willing to commit to group occupational therapy 2x/week for 8 weeks free of charge
* score of at least 4/6 on the short mini mental status exam

Exclusion Criteria:

* less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Fall Risk Factor Management | Baseline, Pre-assessment (8-weeks after baseline), and post-assessment (8-weeks after pre-assessment)
  Self-report 5 scales measuring the ability to manage fall risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Laura Grimm, MS, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No